CLINICAL TRIAL: NCT02665312
Title: CHEmotherapy-induced Cardiotoxicity and Study of risK Factor Correlation in Patients With Colorectal Cancer Receiving Oral or INfusional Fluoropyrimidine Treatment - CHECKPOINT
Brief Title: Cardiotoxicity and Risk Factors in Patients With Colorectal Cancer Receiving Fluoropyrimidine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: CheckPoint
Record Dates: First submitted 2016-01-23; First posted 2016-01-27 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: cardiotoxicity; fluoropyrimidine; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
observational prospective study, designed for patients with colorectal cancer receiving for the first time 5-FU or capecitabine, with or without other chemotherapy combinations.

DETAILED DESCRIPTION:
All patients enrolled will be evaluated for cardiovascular risk factors and, if resulted at cardiovascular risk, they will be submitted to cardiac examination and therapy optimization before starting chemotherapy.

Patients will be evaluated with 12-lead ECG and blood sample for TnI and NT pro-BNP before start chemotherapy and on day 3 of chemotherapy during the first, second and third cycle.

All patients developing cardiovascular events will be submitted to blood sample for TnI, NT-proBNP, hsTnI and cardiac examination.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age ≥ 18 years
* Histologically confirmed adenocarcinoma of colon or rectum (any T, any N, any M) receiving for the first time 5-FU or capecitabine, with or without other chemotherapy combinations

Exclusion Criteria:

* Prior treatment with fluoropyrimidines
* Prior or concurrent chest radiotherapy
* Any prior or concurrent treatment with cardiotoxic drug
* Any serious or uncontrolled cardiovascular disease (defined by the specialist during cardiac examination, see section 6.3.2 for details )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer receiving Oral or INfusional fluoropyrimidine Treatment
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the incidence of cardiovascular events during the first three cycles of therapy with capecitabine or 5-FU | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Leone, MD, Principal Investigator — IRCCS Candiolo
Locations (8):
- Italy (8):
  - Ospedale San Lazzaro - ASL CN 2 Alba Bra, Alba, Cuneo
  - Fondazione del Piemonte per l' Oncologia - IRCCS Candiolo, Candiolo, Turin
  - AO Ordine Mauriziano di Torino, Turin, Turin
  - AOU Città della Salute e della Scienza di Torino - Presidio Molinette - Oncologia Medica 1, Turin, Turin
  - AOU Città della Salute e della Scienza di Torino - Presidio Molinette - Oncologia Medica 2, Turin, Turin
  - Ospedale Cottolengo, Turin, Turin
  - Humanitas Gradenigo, Turin, Turin
  - Ospedale San Giovanni Bosco - ASL TO2, Turin, Turin

IPD SHARING:
Plan to Share IPD: Undecided